CLINICAL TRIAL: NCT02042820
Title: Ocular Surface Immune Response in Dry Eye Disease: Analysis of Conjunctival and Peripheral Corneal Immune Cell Alterations by In Vivo Confocal Microscopy and Clinical Correlation
Brief Title: Ocular Surface Immune Response in Dry Eye Disease
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13-149H
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dry Eye Disease: Confocal Imaging - In vivo confocal microscopy (IVCM)
  Ophthalmic Examination:
  * Tear Break Up Time (TBUT)
  * Ocular Surface Disease Index (OSDI)
  * Schirmer's II test
  * Conjunctival staining with lissamine green
  * Corneal staining with fluorescein
  * Conjunctival redness assessment
  Interventions: Other: In vivo confocal microscopy (IVCM)
- Control: Confocal Imaging - In vivo confocal microscopy (IVCM)
  Ophthalmic Examination:
  * TBUT
  * OSDI
  * Schirmer's II test
  * Conjunctival staining with lissamine green
  * Corneal staining with fluorescein
  * Conjunctival redness assessment
  Interventions: Other: In vivo confocal microscopy (IVCM)

INTERVENTIONS:
Other: In vivo confocal microscopy (IVCM) — IVCM is a sensitive tool for detecting dry eye-associated subclinical inflammation.

SUMMARY:
In vivo confocal microscopy (IVCM) is a sensitive imaging tool for detecting dry eye-associated subclinical inflammation. Studies have previously shown that IVCM provides an in vivo metric to measure inflammatory changes in the central cornea. The objective of the current study is to assess inflammatory response changes in the peripheral cornea and the conjunctiva by analyzing epithelial immune cell density and morphology in these areas and then correlating the IVCM findings to clinical signs and symptoms to establish novel objective imaging biomarkers.

ELIGIBILITY:
For Dry Eye Disease Participants

Inclusion Criteria:

* Age >18
* Ability to consent to study
* Symptoms of dry eye disease for at least 6 months, such foreign body sensation, burning, stinging, light sensitivity
* Positive vital dye staining of the cornea
* At least one of the following objective signs: (Schirmer I <10 mm at 5 minutes), decreased (<0.2 mm) tear meniscus, decreased tear breakup time (TBUT) of <10 seconds, positive vital dye staining of the conjunctiva

For Age-Match Controls

Inclusion Criteria:

* Between the ages of 18-89
* The ability to provide informed consent for study inclusion
* Clear, healthy cornea
* Normal tear meniscus (> 0.3 mm)

For Dry Eye Disease Participants

Exclusion Criteria:

* History of contact lens wear in the past 3 months
* History of ocular surgery in the past 6 months
* Active ocular allergies
* History of ocular infection in the past 3 months
* History of diabetes
* History of topical or systemic anti-inflammatory therapy in the past 1 month

For Age-Match Controls

Exclusion Criteria:

* History of ocular or eyelid surgery within the past 12 months
* History of herpetic or other infectious keratitis or other inflammatory eye disease
* History of any other acute ocular disease
* Current use of topical medications (not including artificial tears)
* Current use of contact lenses
* History of ocular carcinoma or any recent ocular topical chemotherapy or radiotherapy
* History of cancer elsewhere in the body which is currently under systemic chemotherapy
* Current glaucoma disease requiring use of glaucoma drops
* History of Diabetes mellitus
* Current diagnosis of dry eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with and without Dry Eye Disease
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Peripheral Corneal Immune cell Status by IVCM | Visit 1
  Peripheral Corneal Immune cell Status by IVCM • Density of dendritic immune cells • Density of non-dendritic immune cells • Morphology of immune cells
Bulbar conjunctival immune cell Status by IVCM | Visit 1
  Bulbar conjunctival immune cell Status by IVCM • Density of dendritic immune cells • Density of non-dendritic immune cells • Morphology of immune cells

SECONDARY OUTCOMES:
Clinical Parameter: Ocular Surface Disease Index (OSDI) | Visit 1
Clinical Parameter: Schirmer's II test | Visit 1
Clinical Parameter: Conjunctival staining with lissamine green | Visit 1
Clinical Parameter: Corneal staining with fluorescein | Visit 1
Clinical Parameter: Tear Break Up Time (TBUT) | Visit 1
Clinical Parameter: Conjunctival redness | Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — MEEI
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States